## OFFICIAL TITLE OF THE STUDY

Investigation of The Effects of Lumbopelvic Rhythm on Postural Control, Daily Living Activities and Quality of Life in Adolescent Individuals with Idiopathic Scoliosis

## **NCT NUMBER**

NCT Number: Not yet assigned

**DOCUMENT DATE:** 

23 January 2026

(For Individuals with Adolescent Idiopathic Scoliosis)

Dear Participant,

This research, titled "Investigation of the Effect of Lumbopelvic Rhythm and Postural Control on Daily Living Activities and Quality of Life in Adolescent Idiopathic Scoliosis," is being conducted at Hacettepe University Faculty of Physical Therapy and Rehabilitation. We encourage you to participate in this research. However, please note that you are free to participate or not. Participation in this study is voluntary. Before you make your decision, we would like to inform you about the research. After reading and understanding this information, please sign the form if you wish to participate in the research. The reason we want to conduct this research is to examine the movement characteristics of the spine, and especially the lumbar region, in some daily living activities (walking, sitting and standing in a chair) in individuals diagnosed with Adolescent Idiopathic Scoliosis (AIS), to compare them with individuals without this disease, and to reveal possible differences. Your participation in this study, which will be conducted at the Department of Physiotherapy and Rehabilitation, Faculty of Physical Therapy, Hacettepe University, is crucial for the success of the research.

The assessments consist of four parts. First, information such as your age, height, weight, and pain assessment will be collected. Secondly, a 22-question questionnaire assessing quality of life will be administered. Please indicate your answer by marking or writing the option that best suits you. Thirdly, movements in the spine and hips during activities such as bending forward and straightening, bending and straightening to the side, turning the torso to both sides, walking, and getting up from a chair will be evaluated. During this evaluation, five movement-sensing systems, approximately the size of a matchbox, will be placed on the spine (3 on the neck, back, and lumbar region) and on each leg (2 on each leg) using double-sided tape. This system has no effect on the body; it only determines the position of your body parts during the movements. Fourthly, a balance assessment will be conducted. This assessment will be performed on a fixed plate on the floor. Your ability to stand balanced and stable on both open and closed eyes, and on hard and soft surfaces, will be determined. The system has no effect on you. All these assessments will be conducted on the same day and will take approximately 1 hour to complete. The assessments will be carried out in the Movement Analysis Laboratory of the Faculty of Physical Therapy and Rehabilitation.

If you agree to participate in the research, you will be evaluated by the research supervisor, Prof. Dr. Semra TOPUZ, or Specialist Physiotherapist Cem SAMUT, and the results will be recorded. If deemed suitable as a result of the evaluation, you will be included in this study. No fee will be charged for your participation in this study. You will not receive any additional payment for participating in the study.

Your medical information will be kept confidential, but it may be reviewed by the officials overseeing the quality of the study, ethics committees, or official authorities if necessary. You may refuse to participate in this study. Participation in this research is entirely voluntary, and if you refuse, there will be no change in the treatment you receive. You also have the right to withdraw your consent at any stage of the study. (Participant/Patient's Statement) Dear Specialist I was informed by Physiotherapist Cem SAMUT that a research project would be conducted at Hacettepe University, Faculty of Physical Therapy, Department of Physiotherapy and Rehabilitation, and I was subsequently invited to participate in this research.

If I participate in this research, I believe that the confidentiality of my personal information, which should remain between me and the researchers, will be treated with great care and

respect during the research. I have been given sufficient assurance that my personal information will be carefully protected during the use of the research results for educational and scientific purposes.

I may withdraw from the research without giving any reason. Furthermore, I may be excluded from the research by the researcher, provided that my medical condition is not harmed in any way.

I do not assume any financial responsibility for the expenses incurred for the research. I will not receive any payment.

I have been given the necessary assurance that all necessary medical interventions will be provided in the event of any health problems arising directly or indirectly from the research. (I will not incur any financial burden related to these medical interventions either).

I understand that if I encounter a health problem during the research, I can contact Prof. Dr. Semra TOPUZ at 0 312 305 1576 extension: 127 (work) or 0505 580 05 90 (mobile) and Specialist Physiotherapist Cem SAMUT at 0546 500 95 96 or via the Hacettepe University Faculty of Physical Therapy, Department of Physiotherapy and Rehabilitation at any time.

I am not obligated to participate in this research and I may choose not to. I have not been subjected to any coercive behavior regarding my participation. I also understand that if I refuse to participate, this will not negatively impact my medical care or my relationship with the researcher.

I have fully understood all explanations given to me. After a period of independent consideration, I have decided to participate as a "participant" in this research project. I accept this invitation with great pleasure and willingly. I will be given a copy of this signed form.

## Dear Participant,

This research, titled "Investigation of the Effect of Lumbopelvic Rhythm and Postural Control on Activities of Daily Living and Quality of Life in Adolescent Idiopathic Scoliosis," is being conducted at Hacettepe University Faculty of Physical Therapy and Rehabilitation.

We recommend your participation in this research. However, please note that you are free to participate or not. Participation in this study is voluntary. Before you make your decision, we would like to inform you about the research. After reading and understanding this information, if you wish to participate in the research, please sign the form.

The reason we want to conduct this research is to examine the movement characteristics of the spine, and especially the lumbar region, in individuals diagnosed with Adolescent Idiopathic Scoliosis (AIS) during certain daily activities (walking, sitting and standing), to compare them with individuals without this disease, and to reveal any potential differences. Your participation in this study, which will be conducted at the Department of Physiotherapy and Rehabilitation, Faculty of Physical Therapy, Hacettepe University, is important for the success of the research.

The assessment consists of 4 parts. First, information such as your age, height, weight, and pain assessment will be collected. In the second stage, the movements of the spine and hips during activities such as bending forward and straightening, bending and straightening to the side, turning the torso to both sides, walking, and standing up from a chair will be evaluated. During this evaluation, 5 movement-sensing systems, approximately the size of a matchbox, will be placed on the spine (3 on the neck, back, and lumbar region) and on each leg (2 on each leg) using double-sided tape. This system has no effect on the body; it only determines the position of your body parts during movements. In the third stage, a balance assessment will be conducted. This assessment will be performed on a stationary plate on the floor. Your ability to maintain balance and stability on both hard and soft surfaces, with your eyes open and closed, will be determined. The system has no effect on you. All these assessments will be conducted on the same day and will take approximately one hour to complete. The assessments will be carried out in the Movement Analysis Laboratory of the Faculty of Physical Therapy and Rehabilitation. If you agree to participate in the research, you will be evaluated by the research director, Prof. Dr. Semra TOPUZ, or a researcher she designates, and the results will be recorded. If deemed suitable as a result of the evaluation, you will be included in this study.

If you agree to participate in the research, you will be evaluated by the research director, Prof. Dr. Semra TOPUZ, or Specialist Physiotherapist Cem SAMUT, and the results will be recorded. If deemed suitable as a result of the evaluation, you will be included in this study.

You will not be charged any fee for participating in this study. You will not receive any additional payment for participating in the study.

Your medical information will be kept confidential, but may be reviewed by the study's quality control officers, ethics committees, or governmental authorities if necessary.

You may refuse to participate in this study. Participation in this research is entirely voluntary, and refusal will not result in any change to your treatment. You also have the right to withdraw your consent at any stage of the study.

(Participant/Patient's Statement)

I was informed by Specialist Physiotherapist Cem SAMUT that a research project would be conducted at Hacettepe University, Faculty of Physical Therapy, Department of Physiotherapy and Rehabilitation, and I was given the above information regarding this research. Following this information, I was invited to participate in this research.

If I participate in this research, I believe that the confidentiality of my personal information, which should remain between me and the researchers, will be treated with great care and respect during the research. I have been given sufficient assurance that my personal information will be carefully protected during the use of the research results for educational and scientific purposes.

I can withdraw from the research without giving any reason. Furthermore, I can be excluded from the research by the researcher, provided that my medical condition is not harmed in any way.

I do not assume any financial responsibility for the expenses incurred for the research. I will not receive any payment.

I have been given the necessary assurance that all necessary medical intervention will be provided in the event of any health problems arising from the research, whether directly or indirectly. (I will not incur any financial burden regarding these medical interventions.)

I understand that if I encounter a health problem during the research, I can contact Prof. Dr. Semra TOPUZ at 0 312 305 1576 extension: 127 (work) or 0505 580 05 90 (mobile), and Specialist Physiotherapist Cem SAMUT at 0546 500 95 96, or via the Hacettepe University Faculty of Physical Therapy, Department of Physiotherapy and Rehabilitation at any time.

I am not obligated to participate in this research and I may choose not to. I have not encountered any coercive behavior regarding my participation in the research. I also understand that if I refuse to participate, this will not negatively affect my medical care or my relationship with the researcher.

I have fully understood all explanations given to me. After a period of independent consideration, I have decided to participate as a "participant" in the aforementioned research project. I accept this invitation with great pleasure and willingness.

A copy of this signed form will be given to me.